CLINICAL TRIAL: NCT04089644
Title: Physician-Directed vs Computer-Assisted Norepinephrine Administration in Patients Undergoing Major Abdominal Surgery: A Randomized Controlled Trial
Brief Title: Manual vs Closed-loop Control of Mean Arterial Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Collaborators: University of California, Los Angeles (Other); University of California, Irvine (Other); Bicetre Hospital (Other)
Responsible Party: Principal Investigator, Alexandre Joosten, MD PhD, Principal Investigator, Erasme University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P2019/347
Record Dates: First submitted 2019-09-12; First posted 2019-09-13 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Intervention Model Description: Single center prospective randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- manual group (Active Comparator): Hypotension will be corrected by manual infusion of norepinephrine
  Interventions: Device: Manual adjustment
- closed-loop group (Experimental): Hypotension will be corrected by closed-loop control of norepinephrine infusion
  Interventions: Device: closed-loop system

INTERVENTIONS:
Device: closed-loop system — Hypotension will be corrected by an automated system for vasopressor administration.
  Fluids will be given using a goal directed strategy (EV1000 Monitor, Edwards Lifesciences, Irvine, CA, USA)
  Arms: closed-loop group
Device: Manual adjustment — Vasopressor agents will be manually adjusted (standard practice).
  Fluids will be given using a goal directed strategy (EV1000 Monitor, Edwards Lifesciences, Irvine, CA, USA)
  Arms: manual group

SUMMARY:
Intraoperative hypotension can impact patient outcome. Vasopressors are usually used to correct hypotension and ensure adequate organ perfusion.

The investigators have recently developed an automated system (closed-loop system) to titrate vasopressor agents in surgical and intensive care patients.

The purpose of this study is to compare two strategies to correct hypotension based on an individual definition of hypotension (therefore, the target MAP used to define hypotension will differ for each patient (individualized approach):

1. Control group = standard practice ( manually adjusted norepinephrine infusion to correct hypotension and keep MAP within 90% of patient's baseline MAP
2. Intervention group = closed-loop (automated) vasopressor administration system will deliver norepinephrine using feedback from standard operating room hemodynamic monitor (EV1000 Monitor-Flotrac, Edwards Lifesciences, IRVINE, USA) to correct hypotension and keep MAP within 90% of patient's baseline MAP

DETAILED DESCRIPTION:
In order to prevent the known postoperative complications of intraoperative hypotension, vasopressor agents are occasionally used to ensure adequate perfusion. These vasopressors are usually administered as manually adjusted infusions, but this practice requires considerable time and attention.

To overcome this issue, the investigators have developed a closed-loop vasopressor (CLV) controller to potentially correct hypotension more efficiently. After completing extensive in-silico, in-vivo studies and a pilot human trial in a small cohort of 20 patients, the investigators aimed to conduct now a randomized control trial comparing manual vasopressor adjustment versus closed-loop vasopressor adjustment in high risk patients undergoing major abdominal surgeries in order to correct hypotension during surgery

The primary outcome will be the incidence of hypotension (defined as a reduction of > 10% from patient's MAP target, or a allowed tolerance of 10% reduction from patient's baseline MAP). This has been chosen based on the recent study of Emmanuel Futier and colleagues (Effect of Individualized vs Standard Blood Pressure Management Strategies on Postoperative Organ Dysfunction Among High-Risk Patients Undergoing Major Surgery: A Randomized Clinical Trial. JAMA. 2017 Oct 10;318(14):1346-1357), even if it was originally done with systolic blood pressure

Participants in both groups will receive standard patient care in that in no way will their anesthetic or surgical procedure will be altered as part of the study, with the exception of vasopressor administration.

Fluids will be standardized in both groups and will be given as a continuous baseline infusion of 3 ml/kg/h (balanced crystalloid solution) and additional fluid boluses (mini fluid challenges of 100 ml) as a goal directed fluid therapy strategy to maintain stroke volume variation < 13%. The only difference is the way norepinephrine is delivered to the patient (manual versus closed-loop assisted)

ELIGIBILITY:
Inclusion Criteria:

* High-risk adult patients undergoing major abdominal surgeries requiring an advanced cardiac output monitoring device (EV1000-Edwards LifeSciences, Irvine, USA) and a tight blood pressure control

Exclusion Criteria:

* Atrial Fibrillation
* Severe Arythmia

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Percentage of case Time in hypotension (MAP < 90% of the chosen MAP target). | At postoperative day 1
  Undertreatment. Percentage of time during surgery in hypotension. The MAP used to define hypotension will differ for each patient (individualized approach)

SECONDARY OUTCOMES:
Percentage of case time in hypotension (MAP < 65 mmHg) | during surgery
  Percentage of time during surgery in hypotension using the population target usually admitted and used in clinical studies (MAP < 65 mmHg)
Percentage of case time in target (MAP +/- 10 mmHg) of the chosen MAP target | during surgery
  Percentage of time during surgery with a MAP +/- 10 mmHg of the chosen MAP target.
Amount of vasopressors received | during surgery
  Amount of vasopressors received
Uretral perfusion index during surgery | during surgery
  Mean Uretral perfusion index during surgery using the novel IKORUS urinary catheter recently available on the market
Uretral perfusion index during the first 15 minutes of the surgery | during surgery
  Mean Uretral perfusion index during the first 15 minutes of the surgery
Uretral perfusion index during the last 15 minutes of the surgery | during surgery
  Mean Uretral perfusion index during the last 15 minutes of the surgery
Cardiac index during surgery | during surgery
  Mean cardiac index during surgery
Stroke volume index during surgery | during surgery
  Mean Stroke volume index during surgery
Stroke volume variation during surgery | during surgery
  Mean Stroke volume variation during surgery
Amount of fluid received during surgery | during surgery
  Amount of fluid received during surgery
Net fluid balance during surgery | during surgery
  Net fluid balance during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Joosten, MD PhD, Principal Investigator — ERASME
Locations (1):
- Erasme Hospital, Brussels, Brussel-hoofdstad, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Joosten A, Chirnoaga D, Van der Linden P, Barvais L, Alexander B, Duranteau J, Vincent JL, Cannesson M, Rinehart J. Automated closed-loop versus manually controlled norepinephrine infusion in patients undergoing intermediate- to high-risk abdominal surgery: a randomised controlled trial. Br J Anaesth. 2021 Jan;126(1):210-218. doi: 10.1016/j.bja.2020.08.051. Epub 2020 Oct 8. PMID 33041014